CLINICAL TRIAL: NCT04052360
Title: A Single-center, Double-blind, Placebo-controlled, Randomized Study to Investigate the Tolerability, Safety, Pharmacokinetics, and Pharmacodynamics After Single-dose Administration of 4 mg Cenerimod in Healthy Japanese and Caucasian Subjects
Brief Title: Single Oral Dose of 4 mg Cenerimod in Healthy Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID-064-104
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2020-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — cenerimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cenerimod / ACT-334441 (Experimental)
  Interventions: Drug: Cenerimod
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Cenerimod — A single oral dose of 4 mg cenerimod will be administered as a film-coated tablet in the morning of Day 1 under fasted conditions.
  Other Names: ACT-334441
  Arms: Cenerimod / ACT-334441
Drug: Matching Placebo — A single oral dose of matching placebo will be administered as a film-coated tablet in the morning of Day 1 under fasted conditions.
  Arms: Matching Placebo

SUMMARY:
This study is for research purposes only and is not intended to treat any medical condition. The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of cenerimod following a single dose in healthy Japanese and Caucasian participants. Pharmacokinetics is the study of the absorption and breakdown of the study drug in the body. Pharmacodynamics is the study of the effect of the study drug on the body. There will be 2 groups in the study. 10 Japanese participants in one group and 10 Caucasian participants in the other group.

The duration of participation in this study is approximately 75 days from screening to the end of study visit. A screening visit is required within 21 days prior to the start of the study to determine whether the volunteer qualifies and is willing to participate in this research study. This study requires in-patient stay in the research clinic of 4 days (3 nights) followed by outpatient visits and an end of study visit 3 to 5 days after the day 49 outpatient visit.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure.
* Body mass index of 18.0 to 28.0 kg/m^2 (inclusive) at the screening.
* Ability to communicate well with the investigator, in a language understandable to the subject, and to understand and comply with the requirements of the study.
* No clinically relevant findings on the physical examination at screening.
* Systolic blood pressure 100 to 145 mmHg, diastolic blood pressure 50 to 90 mmHg, and pulse rate 55 to 90 bpm (inclusive), measured on the same arm, after 5 min in the supine position at screening and on admission.
* 12-lead ECG without clinically relevant abnormalities, measured after 5 min in the supine position at Screening and on admission.
* No clinically relevant findings in clinical laboratory tests (hematology, clinical chemistry, and urinalysis) at screening and on admission.
* Negative results from urine drug screen and breath alcohol tests at screening and on admission.
* Subjects must be of Caucasian or Japanese ethnicity.

Exclusion Criteria:

* Previous exposure to cenerimod.
* Known hypersensitivity or allergy to natural rubber latex, to or any of the excipients.
* History of major medical or surgical disorders which are likely to interfere with the absorption, distribution, metabolism, or excretion of the study treatment (appendectomy and herniotomy allowed, cholecystectomy not allowed).
* Acute, ongoing, recurrent, or chronic systemic disease able to interfere with the evaluation.
* Clinically relevant history of fainting, collapse, syncope, orthostatic hypotension, or vasovagal reactions.
* Lymphopenia (less than 1.0 x 10^9 cells/L) at screening and on admission.
* Familial history of sick-sinus syndrome.
* Any cardiac condition or illness (including Electrocardiogram (ECG) abnormalities with a potential to increase the cardiac risk.
* Familial history of sick-sinus syndrome.
* Any recent immunosuppressive treatment.
* History or clinical evidence of alcoholism or drug abuse.
* Excessive caffeine consumption, defined as 800 mg or more per day at screening.
* Nicotine consumption within 3 months prior to screening and inability to refrain from nicotine consumption.
* Previous treatment with any prescribed medications (including vaccines) or over-the-counter (OTC) medications (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals).
* Viral, fungal, bacterial or protozoal infection and / or serology.
* Legal incapacity or limited legal capacity at screening.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-11-02 (Actual)

PRIMARY OUTCOMES:
The area under the plasma concentration-time curve (AUC) for cenerimod | From Day 1 to Day 49
  The plasma PK parameter of cenerimod will be derived by non-compartmental analysis of plasma concentration-time profiles.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) for cenerimod | From Day 1 to Day 49
  The plasma PK parameter of cenerimod will be derived by non-compartmental analysis of plasma concentration-time profiles.
Time to reach the maximum plasma concentration (tmax) for cenerimod | From Day 1 to Day 49
  The plasma PK parameter of cenerimod will be derived by non-compartmental analysis of plasma concentration-time profiles.
Terminal half-life [t(1/2)] of cenerimod | From Day 1 to Day 49
  The plasma PK parameter of cenerimod will be derived by non-compartmental analysis of plasma concentration-time profiles.
Lymphocyte count | Day 1, Day 3, Day 6, Day 9, Day 12, Day 15, Day 18, Day 21, Day 28, Day 35, Day 42 and Day 49
  The lymphocyte count will be used as a measure of immunomodulation (a change in the body's immune system).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (1):
- Anaheim Clinical Trials, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No